CLINICAL TRIAL: NCT06701851
Title: Corrélats Neuronaux Des Accès de Mouvements Anormaux Paroxystiques Liées Aux Dyskinésies Paroxystiques kinésigéniques Secondaires à Une Mutation du Gene PRRT2 - Recherche Ancillaire de L'étude AMEDYST " Dont Vous êtes l'Investigateur Principal
Brief Title: Neural Correlates of Movement Disorders Associated With PRRT2 Related Paroxysmal Kinesigenic Dyskinesia - an Ancillary Study of AMEDYST Research
Acronym: TRIGGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C22-09; 022-A02824-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Dyskinesia
Keywords: dyskinesia; voluntary movements; cerebellum; basal ganglia; cortex; fMRI; EEG
MeSH Terms: conditions — Chorea; Dyskinesias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): We will conduct a study using functional MRI and EEG in this subgroup of at least 1 patient(s) with a PRRT2 mutation capable of triggering paroxysmal dyskinesia episodes. We will analyze of the activation of regions involved in the occurrence of abnormal movements during the prodromal phase, during which the acquisition is not affected by movements. We will also investigate the regions involved in judging control over action during phases where abnormal movements may occur before and after the dyskinetic episode.
  Thus, each subject will serve as their own control across different conditions of the experimental paradigm.
  Interventions: Behavioral: Voluntary and involuntary conditions

INTERVENTIONS:
Behavioral: Voluntary and involuntary conditions — An task fMRI/EEG acquisition during the prodromal phase preceding the episode of abnormal movements.
  A task fMRI/EEG acquisition the episode of abnormal movements A task fMRI/EEG acquisition when the subject voluntary mimics the sequence of events (prdrosomal phase + episode of dyskinesia)

SUMMARY:
The main objective of this study is to investigate in real-time the neuronal correlates of paroxysmal dyskinesia episodes related to the PRRT2 mutation within this subgroup of patients (who can control paroxysmal dyskinesia episodes), and more specifically, the pathological role of the reciprocal influence between the striatum and the cerebellum in paroxysmal dyskinesia episodes.

DETAILED DESCRIPTION:
We propose to conduct a study using functional MRI and EEG in this subgroup of patients with the PRRT2 mutation capable of triggering paroxysmal dyskinesia episodes. For both modalities, we aim to perform an analysis of the activation of regions involved in the occurrence of abnormal movements during the prodromal phase when the acquisition is not affected by movements. Using these techniques, we will also investigate the regions involved in judging control over action during phases where abnormal movements may occur before the episode (when the system is excitable) and when it is no longer possible during the refractory period (when the system is no longer excitable). Additionally, we plan to conduct a targeted analysis of functional connectivity in the striato-cerebellar pathway before the episodes (when the system is excitable) and after the episodes during the refractory period (when it is no longer excitable).

Our hypotheses are as follows: 1) there is a relationship between the cerebellum, the basal ganglia and the cortex implicated in the abnormal movements associated with the PRRT2 mutation; 2) the frontal or prefrontal cortex, the cerebellum and basal ganglia are involved in the inhibition of unwanted movements; 3) there is a distortion in the sense of control over action related to paroxysmal dyskinesia episodes.

ELIGIBILITY:
Inclusion Criteria:

Male or female Individuals with dystonic disease carrying a PRRT2 mutation and demonstrating the ability to control paroxysmal dyskinesia episodes.

Affiliated with a health insurance system or a beneficiary of such a system. Individuals aged 18 to 75 years. Signature of informed consent

Exclusion Criteria:

Individuals under guardianship. Individuals not residing in France. Individuals unable to comply with protocol constraints (compliance with visit schedules and ability to perform required tasks).

Individuals undergoing an exclusion period for another research study. Contraindications to MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
BOLD signal amplitude | Visit 1 to 5
EEG signal amplitude | Visit 6 to 10

SECONDARY OUTCOMES:
Perception of control over an movement | Visit 11 to Visit 14 (optional)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Cerveau de la Moelle Epinière ICM, Hôpital Pitié Salpêtrière,, Paris, France

IPD SHARING:
Plan to Share IPD: No
Due to ethical policies